CLINICAL TRIAL: NCT06582550
Title: Effectiveness of Audiovisual Versus Written Postoperative Instructions for Patients Undergoing Minor Hand Procedures: a Prospective Controlled Trial
Brief Title: Effectiveness of Audiovisual Versus Written Postoperative Instructions for Patients Undergoing Minor Hand Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Stephanie Thibaudeau, Assistant Professor of Plastic Surgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-10990
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Carpal Tunnel Syndrome; Hand Cyst Ganglion; Trigger Finger
MeSH Terms: conditions — Carpal Tunnel Syndrome; Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: Note that the surgical intervention is the same in both study arms. The comparison is in regards to the post-operative instructions with the aim of quality improvement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Audiovisual Instruction Group (Experimental): Patients who require a hand surgery presenting to the clinic will be divided randomly; each participant is assigned by opening a prepared envelope with a dedicated group randomly, if the patient is assigned to group 1, they will receive standard printed instructions regarding their expected postoperative care, but if the patient is assigned to group 2, they will be provided with a barcode to scan to view audiovisual instructions regarding their post-operative course
  Interventions: Procedure: Minor Hand Procedure
- Written Instruction Group (Active Comparator): Patients who require a hand surgery presenting to the clinic will be divided randomly; each participant is assigned by opening a prepared envelope with a dedicated group randomly, if the patient is assigned to group 1, they will receive standard printed instructions regarding their expected postoperative care, but if the patient is assigned to group 2, they will be provided with a barcode to scan to view audiovisual instructions regarding their post-operative course
  Interventions: Procedure: Minor Hand Procedure

INTERVENTIONS:
Procedure: Minor Hand Procedure — Unilateral minor hand procedure (carpal tunnel release, trigger finger A1 pulley release, lesion excision)

SUMMARY:
The utility and effectiveness of video-based instructions (VBI) versus standard written instructions was not previously investigated in hand surgery; thus, the objective of this study is to evaluate the effectiveness of audiovisual instruction as compared to regular verbal instructions given to patients undergoing common hand procedures, including instruction recall and compliance, patient education, patient satisfaction with the information given, patient satisfaction with operative experience.

DETAILED DESCRIPTION:
Outcomes of hand surgery are greatly dependent on factors outside the operating theater as well. These include patient compliance to preoperative instructions that consist of proper surgical site care, proper positioning, and following occupational therapy protocols. Previous studies have shown that video-based information provide greater patient satisfaction than verbal instructions. Visual information was also reported to decrease patient anxiety regarding the procedure and increases patient education in terms of procedure risks and benefits(1-5). The utility and effectiveness of video-based instructions (VBI) versus standard written instructions was not previously investigated in hand surgery; thus, the objective of this study is to evaluate the effectiveness of audiovisual instruction as compared to regular verbal instructions given to patients undergoing common hand procedures, including instruction recall and compliance, patient education, patient satisfaction with the information given, patient satisfaction with operative experience. The secondary objective is to evaluate if VBI result in better outcomes than standard written instructions.

ELIGIBILITY:
Inclusion Criteria:

Please ensure that ALL items below are satisfied to be included in the study.

* Patient undergoing hand and/or upper extremity surgery with Dr. Thibaudeau
* Patient ≥ 18 years old
* Patient who comprehends instructions provided in English and/or French
* Patient who can navigate the internet to complete an online post-operative questionnaire

Exclusion Criteria:

Please ensure that NONE of the following items are selected to be included in the study.

* Patient presenting with intra-articular, open, or pathological fractures
* Patient presenting with associated tendon or nerve injuries
* Patient receiving definitive surgery ≥21 days after injury
* Patient with previous surgeries/deformity in the hand
* Patient with pre-existing severe joint disease (rheumatoid arthritis, finger joint stiffness, or non-union)
* Patient with medical contraindications to surgery
* Patient who is unable to comply with rehabilitation
* Patient who is unwilling to be followed up
* Patient with dementia
* Patient with significant mental illness
* Patient who is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-19 (Estimated); Primary Completion 2025-09-19 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction with the operative experience | within 1 week
  Questionnaire to assess patient satisfaction with the operative experience will be distributed within a week in post operative visit
patient instruction recall | within 1 week
  Questionnaire to assess patient instruction recall will be distributed within a week in post operative visit. It consists of 9 questions, the maximum score is 9 and indicates excellent recall.
patient satisfaction with the information given | within 1 week
  Questionnaire to assess patient satisfaction with the information givenwill be distributed within a week in post operative visit
  Overall, are you satisfied with the provided post-operative instructions for your hand surgery? Likert-scale 1-10 (with smile face) Overall, were the provided post-operative instructions for your hand surgery easy to understand? Likert-scale 1-10 (with smile face) Overall, did the provided post-operative instructions for your hand surgery had the appropriate amount of information? Likert-scale 1-10 (with smile face)
patient compliance | within 1 week
  Questionnaire to assess patient instruction compliance will be distributed within a week in post operative visit. It consists of 13 questions, each with a score, with 13 being thre maximum patient compliance.

SECONDARY OUTCOMES:
Nursing staff patient experience | within 3 months
  Nursing staff will be asked to present which patients reached out to clinic number/email with questions and if the instrutions decreased the incidence of such
  Assessed as binomial outcome
  Have you called your surgeon's office post-operatively regarding any unexpected post-operative course? Yes No Unsure
Dash Scores | within 1 week
  Questionnaire to assess patient outcome will be distributed within a week in post operative visit
  Quick dash score
  QuickDASH DISABILITY/SYMPTOM SCORE= (sum of n responses) - 1 x 25, wherenis equal to the number of completed responses.

IPD SHARING:
Plan to Share IPD: Undecided